CLINICAL TRIAL: NCT03803683
Title: mLab App for Improving Uptake of Rapid HIV Self-testing and Linking Youth to Care
Brief Title: Improving Health Outcomes in Young Cisgender Men and Transgender Women (mLab App)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rebecca Schnall, RN, MPH, PhD (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Rebecca Schnall, RN, MPH, PhD, Mary Dickey Lindsay Associate Professor of Disease Prevention and Health Promotion, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AAAR8760; R01MH118151 (NIH)
Record Dates: First submitted 2018-09-02; First posted 2019-01-14 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: HIV Infections
Keywords: mLab; HIV prevention
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- mLab App Intervention (Experimental): Youth randomized to the intervention arm (arm 1) will be provided with the mLab App, 2 OraQuick tests (including the package insert), and a box of condoms to take home at baseline. They will receive 2 more OraQuick tests at their 6 month visit. At their baseline appointment, youth will also be sent an email or text with links to mobile-optimized online prevention information, including PrEP and HIV testing information that is found on the CDC website. They will also receive a study information card listing the Columbia University School of Nursing / Lurie Children's study teams' contact information.
  Interventions: Device: mLab App; Behavioral: HIV Prevention Information; Device: HIV Home Tests
- Standard of Care HIV Information Control Arm (Active Comparator): Youth randomized to the Standard of Care HIV information control arm (arm 2) will receive standard-of-care HIV/STI testing-related risk reduction counseling, a box of condoms, PrEP assessment, and referral information for clinics that provide PrEP during their first visit. Youth randomized to the standard of care will be sent an email with links to mobile-optimized online prevention information, including pre-exposure prophylaxis (PrEP) and HIV testing information that is found on the CDC website.They will also receive a study information card listing the Columbia University School of Nursing / Lurie Children's study teams' contact information.
  Interventions: Behavioral: HIV Prevention Information
- HIV Home Tests (Active Comparator): Youth randomized to the HIV home testing arm (arm 3) will be provided with the 2 OraQuick tests (including the package insert), and a box of condoms to take home at baseline. They will receive 2 more OraQuick tests at the 6 month visit. At their baseline appointment, youth will also be sent an email or text with links to mobile-optimized online prevention information, including PrEP and HIV testing information that is found on the CDC website. They will also receive a study information card listing the Columbia University School of Nursing / Lurie Children's study teams' contact information.
  Interventions: Behavioral: HIV Prevention Information; Device: HIV Home Tests

INTERVENTIONS:
Device: mLab App — The mLab App is a web application that uses an image processing algorithm to interpret the results of the OraQuick® In-Home HIV Test.
  Arms: mLab App Intervention
Behavioral: HIV Prevention Information — Youth randomized to the standard of care will be sent an email with links to mobile-optimized online prevention information, including PrEP and HIV testing information that is found on the Centers for Disease Control and Prevention (CDC) website.
Device: HIV Home Tests — Youth randomized into this arm will receive OraQuick® In-Home HIV Test.
  Arms: HIV Home Tests; mLab App Intervention

SUMMARY:
The mLab App combines HIV prevention information with push notifications/reminders to complete HIV testing and an automated image processing feature to provide real-time feedback on home-based HIV test results. Theoretically-guided by the Health Information Technology Usability Evaluation Model (Health-ITUEM), the proposed project will refine and test a next-generation diagnostic intervention delivered on a mobile platform to improve HIV testing and linkage-to-care outcomes among youth living with and at-risk for HIV. Given the pervasiveness, low cost, and convenience of mobile technology, the investigators hope that the App can help achieve the goals of the National HIV/AIDS Strategy in the US by increasing the number of persons living with HIV who know their serostatus, decreasing HIV-related disparities, and ultimately reducing the risk of HIV transmission and acquisition.

DETAILED DESCRIPTION:
The number of youth living with human immunodeficiency virus (HIV) continues to rise, and they are disproportionately represented at each stage of the care continuum. Most relevant to this study, it is estimated that less than half of HIV-infected youth in the United States (US) have been diagnosed with HIV, and acquired immunodeficiency syndrome (AIDS)-related deaths among youth have increased over the past decade despite decreased death rates among all other age groups, pointing to the urgent need for increased testing among youth.

Black and Latino youth are at increased risk of poor HIV-related outcomes and have disparate testing rates as compared to White youth. Mobile Health (mHealth) technology is a powerful and relevant tool which represents a promising approach for improving outcomes among youth living with HIV. Youth are avid adopters and heavy users of smartphones and digital technologies, and these technologies offer opportunities to tailor interventions to developmental stages and personal needs. Importantly, these technologies are capable of delivering interventions in real-time and in ecologic settings. This creates an opportunity to remotely reach youth through mobile and connected health approaches to strengthen their HIV care continuum engagement and treatment outcomes. In response, the investigators have developed the mLab App, an innovative mobile and connected technology that combines HIV prevention information with push notifications/reminders to complete HIV testing and an automated image processing feature to provide accessible, objective, secure, and real-time feedback on home-based OraQuick (lateral flow assay) HIV test results. The mLab App also contains an innovative automated data collection and a results reporting feature. Findings from the investigators' preliminary work in New York City indicate that youth perceive the mLab App as useful, easy to use, and effective at improving health outcomes and intend to use the technology. Furthermore, preliminary work in Africa support the sensitivity and specificity of the imaging algorithm for interpreting lateral flow assay results.

The investigators will conduct a careful, iterative process of technology refinement based on input from end users, experts, and the youth advisory board. The investigators will then enroll 525 high-risk youth (age 18-29 years) in a 12-month randomized controlled trial (RCT) to assess differences in HIV testing rates and linkage to care between three arms the intervention arm, the standard of care-HIV information control arm, and the HIV home test arm. Finally, the investigators will analyze paradata, defined as auxiliary data that capture details about the process of interaction with the technology, to understand the effect of user engagement of the mLab App on improving HIV testing rates and linkage to care. Interventions delivered through mHealth technology represent a promising approach for improving outcomes among youth.

ELIGIBILITY:
Inclusion Criteria:

* Birth sex male of any current gender identification;
* Understand and read English
* Substantial risk for acquiring HIV infection per CDC guidance (e.g.,YMSM or YTGW and recent anal sex with men)
* Smartphone ownership
* Self-report being HIV-negative or unknown status
* Understand the limitations of the OraQuick test and the mLab App
* Not having been tested for HIV in the past 6 months (e.g., therefore being somewhat outside of the current CDC testing recommendations for high-risk populations)
* Not currently taking PrEP
* Receive a non-reactive result on the rapid HIV test at the Baseline visit

Exclusion Criteria:

* Persons who have a known diagnosis of HIV
* Persons for whom the investigators determine that participation may be detrimental to the participant or to the study (e.g., severe cognitive deficit).

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 525 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, RN, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Lurie Children's Hospital, Chicago, Illinois
  - Columbia University School of Nursing, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schnall R, Scherr TF, Kuhns LM, Janulis P, Jia H, Wood OR, Almodovar M, Garofalo R. Efficacy of the mLab App: a randomized clinical trial for increasing HIV testing uptake using mobile technology. J Am Med Inform Assoc. 2025 Feb 1;32(2):275-284. doi: 10.1093/jamia/ocae261. PMID 39560363
- [Derived] Wood OR, Garofalo R, Kuhns LM, Scherr TF, Zetina APM, Rodriguez RG, Nash N, Cervantes M, Schnall R. A randomized controlled trial of an mHealth intervention for increasing access to HIV testing and care among young cisgender men and transgender women: the mLab App study protocol. BMC Public Health. 2021 Oct 29;21(1):1959. doi: 10.1186/s12889-021-12015-w. PMID 34715833

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 525 participants enrolled, however 523 were randomized as two participants withdrew prior to randomization.
Period: Overall Study
Arm/Group | mLab App Intervention | Standard of Care HIV Information Control Arm | HIV Home Tests
Started | 211 | 208 | 104
Completed | 161 | 189 | 88
Not Completed | 50 | 19 | 16
Not completed — Lost to Follow-up | 41 | 18 | 12
Not completed — Withdrawal by Subject | 9 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mLab App Intervention | Standard of Care HIV Information Control Arm | HIV Home Tests | Total
Number analyzed (Participants) | 211 | 208 | 104 | 523
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (3.23) | 23.9 (3.34) | 24.3 (3.28) | 24.1 (3.28)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 186 | 193 | 96 | 475
  Trans Feminine | 7 | 2 | 4 | 13
  Genderqueer | 7 | 0 | 2 | 9
  Non-binary | 9 | 13 | 1 | 23
  Other | 2 | 0 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 73 | 61 | 26 | 160
  Not Hispanic or Latino | 137 | 147 | 77 | 361
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 2 | 4 | 1 | 7
  Asian or Asian American | 25 | 31 | 11 | 67
  Black or African-American | 22 | 19 | 6 | 47
  Hispanic or Latino/Latinx | 5 | 6 | 1 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  White or Caucasian | 123 | 118 | 62 | 303
  Multiracial | 21 | 13 | 15 | 49
  Something else | 12 | 17 | 6 | 35
  Unknown/Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 211 | 208 | 104 | 523
Sexual Orientation [Count of Participants; unit: Participants]
  Bisexual | 36 | 24 | 12 | 72
  Gay/homosexual | 142 | 156 | 82 | 380
  Queer | 25 | 27 | 5 | 57
  Straight/heterosexual | 2 | 1 | 2 | 5
  Other | 6 | 0 | 3 | 9
Any HIV test in the past 6 months [Count of Participants; unit: Participants] | 74 | 60 | 22 | 156

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Youth Tested for HIV
Description: Total number of youth tested for HIV at 6 months
Time Frame: 6 months
Population: 175 in Arm1, 189 in Arm 2, and 94 in Arm 3 analyzed as this was the number of participants that completed the 6 month visit and from which data was collected.
Measure: Count of Participants; unit: Participants
Arm/Group | mLab App Intervention | Standard of Care HIV Information Control Arm | HIV Home Tests
Number analyzed (Participants) | 175 | 189 | 94
Participants | 154 | 123 | 68

2. Primary Outcome: Total Number of Youth Tested for HIV
Description: Total number of youth tested for HIV at 12 months
Time Frame: 12 months
Population: 161 in Arm1, 189 in Arm 2, and 88 in Arm 3 analyzed as this was the number of participants that completed the 12 month visit and from which data was collected.
Measure: Count of Participants; unit: Participants
Arm/Group | mLab App Intervention | Standard of Care HIV Information Control Arm | HIV Home Tests
Number analyzed (Participants) | 161 | 189 | 88
Participants | 145 | 109 | 64

3. Secondary Outcome: Total Number of HIV Negative/ Positive Results
Description: Total number of HIV negative/ positive results at 6 months
Time Frame: 6 months
Population: 154 in Arm 1, 123 in Arm 2, and 68 in Arm 3 analyzed as this was the number of participants that completed the HIV test and from which data was collected.
Measure: Count of Participants; unit: Participants
Arm/Group | mLab App Intervention | Standard of Care HIV Information Control Arm | HIV Home Tests
Number analyzed (Participants) | 154 | 123 | 68
Participants
  Negative | 154 | 123 | 68
  Positive | 0 | 0 | 0

4. Secondary Outcome: Total Number of HIV Negative/ Positive Results
Description: Total number of HIV negative/ positive results at 12 months
Time Frame: 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mLab App Intervention | Standard of Care HIV Information Control Arm | HIV Home Tests
Number analyzed (Participants) | 161 | 189 | 88
Participants
  Negative | 161 | 189 | 88
  Positive | 0 | 0 | 0

5. Secondary Outcome: Total Number of Youth Who Link to HIV Care Services
Description: Total number of youth who link to HIV care services at 6 months
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | mLab App Intervention | Standard of Care HIV Information Control Arm | HIV Home Tests
Number analyzed (Participants) | 175 | 189 | 94
Participants | 0 | 0 | 0

6. Secondary Outcome: Total Number of Youth Who Link to HIV Care Services
Description: Total number of youth who link to HIV care services at 12 months
Time Frame: 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mLab App Intervention | Standard of Care HIV Information Control Arm | HIV Home Tests
Number analyzed (Participants) | 161 | 189 | 88
Participants | 0 | 0 | 0

7. Secondary Outcome: Number of Sexual Partners in the Past 3 Months
Description: Number of Sexual Partners in the past 3 months collected at the 6 month mark
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: partners
Arm/Group | mLab App Intervention | Standard of Care HIV Information Control Arm | HIV Home Tests
Number analyzed (Participants) | 175 | 189 | 94
partners | 2.12 (3.98) | 1.69 (3.56) | 1.78 (1.90)

8. Secondary Outcome: Number of Sexual Partners in the Past 3 Months
Description: Number of Sexual Partners in the past 3 months collected at the 12 month mark
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: partners
Arm/Group | mLab App Intervention | Standard of Care HIV Information Control Arm | HIV Home Tests
Number analyzed (Participants) | 161 | 189 | 88
partners | 2.24 (4.80) | 2.11 (7.44) | 2.43 (3.57)

9. Secondary Outcome: Number of Condomless Anal Sex Acts
Description: Number of condomless anal sex acts in the past 3 months at 6 months
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: condomless anal sex acts
Arm/Group | mLab App Intervention | Standard of Care HIV Information Control Arm | HIV Home Tests
Number analyzed (Participants) | 175 | 189 | 94
condomless anal sex acts | 7.35 (15.34) | 8.21 (21.67) | 7.56 (9.93)

10. Secondary Outcome: Number of Condomless Anal Sex Acts
Description: Number of condomless anal sex acts in the past 3 months at 12 months
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: condomless anal sex acts
Arm/Group | mLab App Intervention | Standard of Care HIV Information Control Arm | HIV Home Tests
Number analyzed (Participants) | 161 | 189 | 88
condomless anal sex acts | 7.01 (12.15) | 8.33 (15.75) | 8.32 (11.49)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | mLab App Intervention | Standard of Care HIV Information Control Arm | HIV Home Tests
All-Cause Mortality (participants affected / at risk) | 0/211 | 0/208 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/211 | 0/208 | 0/104
Other Adverse Events (participants affected / at risk) | 0/211 | 0/208 | 0/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT03803683/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT03803683/ICF_001.pdf